CLINICAL TRIAL: NCT00371787
Title: Evaluation of the Performance of Non-molded Soft Contact Lenses
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: CIBA VISION (Industry)
Responsible Party: Craig Woods, Research Manager, CCLR
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P/240/06/CV
Record Dates: First submitted 2006-09-01; First posted 2006-09-04 (Estimated); Results first posted 2010-12-13 (Estimated); Last update posted 2011-01-10 (Estimated); Status verified 2011-01

CONDITIONS: Ametropia
MeSH Terms: conditions — Refractive Errors | interventions — Contact Lenses, Hydrophilic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- soft contact lens (Experimental)
  Interventions: Device: Soft contact lens
- non-lens wear (No Intervention): control group

INTERVENTIONS:
Device: Soft contact lens — Soft contact lens
  Other Names: Custom O2Optix
  Arms: soft contact lens

SUMMARY:
To evaluate the performance of the study soft lens for vision, comfort, physiology and lens surface properties.

DETAILED DESCRIPTION:
To evaluate the performance of the study soft lens for vision, comfort, physiology and lens surface properties in a group of participants who present with lens related changes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, good health, age >17yrs, able to wear contact lenses as primary vision correction, able to see well and achieve good fit with study lens, has understood & signed consent form.

Exclusion Criteria:

* Has active ocular disease, uses topical eye medication, wears gas permeable/silicone hydrogel /overnight wear contact lenses, is a participant in another clinical study, is deemed unsuitable for soft contact lens wear.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2006-08; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Desmond Fonn, Principal Investigator — Centre for Contact Lens Research
Locations (1):
- Centre for Contact Lens Research, University of Waterloo,, Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from local communities in Kitchener-Waterloo, Canada between July 2006 and Feb 2007
Pre-assignment Details: 38 participants recruited and screened; 4 withdrew by subject
Groups:
- Treatment Group: soft lens wearers with sign of hypoxia and high prescription
- Control Group: normal non-lens wearers
Period: Overall Study
Arm/Group | Treatment Group | Control Group
Started | 26 | 12
Completed | 23 | 11
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Control Group | Total
Number analyzed (Participants) | 26 | 12 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 12 | 38
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 31.6 (10.75) | 33.25 (6.9) | 32.4 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 8 | 26
  Male | 8 | 4 | 12
Region of Enrollment [Number; unit: participants]
  Canada | 26 | 12 | 38

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: level of vision measured using high contrast acuity chart, higher (more positive)logMAR indicates worse vision.
Time Frame: baseline
Population: Per Protocol. Only the data from participants who completed all study visits were analyzed.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 26 | 12
logMAR | 0.01 (0.09) | -0.07 (0.11)

2. Primary Outcome: Visual Acuity
Description: level of vision measured using high contrast acuity chart, higher (more positive)logMAR indicates worse vision.
Time Frame: 9 month
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 26 | 12
logMAR | 0.01 (0.09) | -0.08 (0.10)

3. Primary Outcome: Neovascularisation
Description: length of the blood vessels entering the superior cornea, higher number means longer blood vessel penetration.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 26 | 12
mm | 0.84 (0.39) | 0.35 (0.16)

4. Primary Outcome: Neovascularization
Description: length of the blood vessels entering the superior cornea, higher number means longer blood vessel penetration.
Time Frame: 9 month
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 26 | 12
mm | 0.63 (0.2) | 0.35 (0.19)

ADVERSE EVENTS:
Arm/Group | Treatment Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/12
Other Adverse Events (participants affected / at risk) | 0/26 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No